CLINICAL TRIAL: NCT00999765
Title: Pilot Study: Mindfulness-Based Cognitive Therapy as a Tool for Prophylactic Mood Stabilizing Therapy in Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: Douglas Mental Health University Institute (Other)
Responsible Party: Principal Investigator, Serge Beaulieu, Serge Beaulieu, Douglas Mental Health University Institute
Other Study IDs: BD-MBCT
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Bipolar Depression; Mindfulness-Based Cognitive Therapy; MBCT; Maintenance; Euthymic; Efficacy; Feasibility
MeSH Terms: conditions — Bipolar Disorder | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bipolar Disorder - stable
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — eight-week (two hours a week) group therapy (8-12 patients per group)

SUMMARY:
The purpose of this study is to evaluate the feasibility and short-term efficacy of MBCT as an add-on (i.e. patients must be stable with their regular mood stabilizing medication) for the maintenance therapy of bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Males or females (>18 years old)
* Bipolar disorder (as per the Structured Clinical Interview for DSM Disorders (SCID)(22)), euthymic state: Complete remission for at least four weeks ((Montgomery and Asberg Rating Scale (MADRS) ≤ 6 and item-1 (depressed mood) = 0 and no suicidal ideations (MADRS(item-10) < 4)
* Must have had at least 3 depressive phases in the last 5 years
* Cooperative and willing to complete all the aspects of the study and especially the 45 minutes of exercise per day
* Must have completed a Secondary V (11th grade) education

Exclusion Criteria:

* Other active psychiatric disorders (as per the SCID)
* Rapid cycling
* Bipolar disorder secondary to a medical condition or substance-induced mood disorder
* Suicidal ideations (MADRS(item 10)>3)
* Active i.e. unstable and/or untreated medical condition
* Substance abuse (defined as per DSM-IV) in the last four weeks
* CBT (No more than four sessions (ever))
* Previous participation in a psychoeducation group within the last 6 months
* Current other psychotherapy (more than once a month)
* Practice of meditation (more than once a month) during the last two years
* Practice of yoga (more than once a week) during the last year
* Previous participation in a MBSR group
* Electroconvulsive Therapy (ECT) within the last three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bipolar Disorder of third-line bipolar disorders program
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
number of weeks in which criteria are meet for a mood episode evaluate with the Longitudinal Interval Follow-up Evaluation (LIFE) | 12 weeks (4 weeks post treatment)

SECONDARY OUTCOMES:
Change in intensity of subsyndromal symptoms of depression on the HAM-D 29 scale | 2, 4, 6, 8 and 12 weeks
Change in intensity of subsyndromal symptoms of depression on the MADRS scale | 2, 4, 6, 8 and 12 weeks
Change in intensity of subsyndromal symptoms of hypomania on the YMRS scale | 2, 4, 6, 8 and 12 weeks
Change id intensity in subsyndromal symptoms of anxiety on the HAM-A scale | 2,4,6,8 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Serge Beaulieu, Ph.D., Principal Investigator — Douglas Mental Health University Institute / McGill
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada